CLINICAL TRIAL: NCT05244460
Title: Droperidol on Prevention of Emesis From Cannabinoid Hyperemesis Syndrome
Brief Title: Droperidol on Prevention of Cannabis Hyperemesis Syndrome
Acronym: DOPE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mercy Health Ohio (Other)
Collaborators: Lake Erie College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-029
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Cannabis Hyperemesis Syndrome
MeSH Terms: conditions — Cannabinoid Hyperemesis Syndrome | interventions — Droperidol; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Patients who receive droperidol 2.5mg intravenous once and diphenhydramine 25mg intravenous once
  Interventions: Drug: Droperidol Injectable Product; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Droperidol Injectable Product — Treatment
  Other Names: Inapsine
Drug: Diphenhydramine — Treatment
  Other Names: Benadryl

SUMMARY:
The purpose of this study is to assess the efficacy of droperidol as a treatment of cannabinoid hyperemesis syndrome.

DETAILED DESCRIPTION:
Patients presenting to the Emergency Department with nausea, vomiting and/or abdominal pain with a significant history of cannabis use and symptoms in a cyclic pattern will be assessed for study inclusion. After given written informed consent, patients will be treated with droperidol and diphenhydramine and symptoms will be assessed using a visual analog scale at time intervals up to 120 minutes. Patient will then be contacted at 24 and 48 hour intervals to assess symptoms on the same scale. This is a multicenter, prospective interventional study with results compared to a historical cohort using haloperidol.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years of age or older and presenting with cannabis hyperemesis syndrome requiring intravenous medication.

Exclusion Criteria:

* any patient with a contraindication to the use of droperidol
* Corrected QT interval on ECG greater than 440 milliseconds for males and greater than 450 milliseconds for females
* any prisoners
* pregnant females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in symptoms after treatment with droperidol and diphenhydramine | Baseline, 30 minutes, 60 minutes and 120 minutes. Then at 24 hours and 48 hours.
  The Visual Analog Scale is a 100-mm patient-reported score measurement used to assess nausea and/or vomiting and/or abdominal pain. Possible scores range from 0 (symptom-free) to 10 (worst possible symptom)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bolotin, MD, Principal Investigator — Mercy Health
Locations (4):
- United States (4):
  - Mercy Health - Austintown, Austintown, Ohio
  - St Elizabeth Boardman Hospital, Boardman, Ohio
  - St. Joseph-Warren Hospital, Warren, Ohio
  - St Elizabeth Youngstown Hospital, Youngstown, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruberto AJ, Sivilotti MLA, Forrester S, Hall AK, Crawford FM, Day AG. Intravenous Haloperidol Versus Ondansetron for Cannabis Hyperemesis Syndrome (HaVOC): A Randomized, Controlled Trial. Ann Emerg Med. 2021 Jun;77(6):613-619. doi: 10.1016/j.annemergmed.2020.08.021. Epub 2020 Nov 5. PMID 33160719
- [Background] Lee C, Greene SL, Wong A. The utility of droperidol in the treatment of cannabinoid hyperemesis syndrome. Clin Toxicol (Phila). 2019 Sep;57(9):773-777. doi: 10.1080/15563650.2018.1564324. Epub 2019 Feb 7. PMID 30729854
- [Background] Hickey JL, Witsil JC, Mycyk MB. Haloperidol for treatment of cannabinoid hyperemesis syndrome. Am J Emerg Med. 2013 Jun;31(6):1003.e5-6. doi: 10.1016/j.ajem.2013.02.021. Epub 2013 Apr 10. PMID 23583118